CLINICAL TRIAL: NCT06709352
Title: Association Between Anti-hypertensive Drugs and Root Caries Among Senior Patients Attending Cairo University Dental Educational Hospital : Analytical Cross-Sectional Study
Brief Title: Effect of Hypertensive Drugs on Root Caries Among Senior Patients in Cairo University
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nuha Abdelrahman Abdelhai Elhaj, Nuha Abdelrahman Abdelhai Elhaj (DDS), Cairo University
Other Study IDs: Root Caries & Drugs
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Root Caries; Antihypertensive Drugs
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: non — non

SUMMARY:
The aim of this analytical cross-sectional study study is to evaluate the prevalence of root caries in senior patients of both genders age of 50 to 70 years old, taking antihypertensive drugs attending the Cairo University Dental Educational Hospital and to consider the association of root caries with antihypertensive drugs. Furthermore, to understand the relationship between risk indicators of root caries and saliva pH that can be a potential etiological factor.

- The main question it aims to answer is: In senior patients attending Cairo University Dental Educational Hospital, what is the prevalence of root caries among patients taking antihypertensive drugs, what are the related risk indicators and how do they correlate with salivary pH?

DETAILED DESCRIPTION:
1. Introduction and Scientific Background:

   Root caries is a condition that commonly affects the senior population worldwide. It's a result of physiological gingival recession with aging that may be greatly exacerbated by poor oral hygiene. (Delphine, S. et al, 2023). In Egypt, caries prevalence is estimated to be (60-70%). (Marwa M.S. Abbass et al,2019).

   In a systematic review, respondents from all nine groups of countries including Egypt, reported that elderly age group (i.e., >60 years old) considered to be most susceptible to developing root caries. (Qutieshat A, 2021). Oral conditions like root caries are known to be caused by a number of systemic factors, one of which is hypertension. Hypertension is a long-term medical condition characterised by elevated blood pressure within the arteries.

   The national estimate for the prevalence of hypertension in Egypt's adult population is 26.3%, making it one of the highest in the world, according to The Egyptian National Hypertension Project (NHP). (Khalafallah, M. et al. 2023). When used as a treatment for hypertension, antihypertensive drugs can have variety of adverse effects on the mouth, including xerostomia and abnormal salivary flow, which leads to dental caries. Also, numerous negative alterations in the oral cavity can be linked to conclusive impact of stimulated saliva on pH.

   (Delphine, S. et al, 2023). Although further investigation is necessary to fully comprehend the connection between antihypertensive medications and dental health, these results imply that using these drugs has an impact on oral health and necessitates maintaining proper oral hygiene.
2. Review of Literature:

   A key element of "Active Ageing" is health. Root caries is one of the main oral public health issues linked to aging. Over the past forty years, there has been a notable decrease in the number of edentulous people and an increase in the number of natural teeth that are still in the oral cavity, according to periodic dental health surveys. Because life expectancy has increased over the past few decades, a significant portion of the population is now older. (S.R. Lingaladinne 2021).

   According to studies, over half the individuals older than 65 years have experienced root caries. It's also suggested that adults who have lived in fluoridated areas throughout most of their lives, including the time of tooth formation, have a lower prevalence of root caries. (Alexandre R. Vieira ,2011)

   Such findings are in line with other studies that estimated that caries prevalence In Egypt was about (60-70%). Egyptian adults proved to be at greater risk of developing caries, with a total prevalence of 86.63%; as compared to children and adolescence, for whom a value of 74% was recorded. (Marwa M.S. Abbass et al,2019).

   Studies have shown that antihypertensive drugs can cause adverse reaction which is defined by the WHO as 'a response to a drug which is noxious and unintended. It occurs at doses normally used in man for the diagnosis, therapy of diseases or for the modification of physiological function. (Delphine, S. et al, 2023).

   These Drugs have the potential to cause conditions such as dental caries, salivary gland disease, ulceration, taste alterations, discolouration of teeth, mucosal pigmentation, white lesions and swellings. These side effects interfere with the patient's normal function and increases the risk of infection, pain and possible tooth loss. Common side effects include dental caries, xerostomia, Altered taste and stomatitis.

   While more research is needed to understand the relationship between antihypertensive drugs and oral health, these findings suggest that taking these medications impacts one's oral health therefore requires good oral hygiene maintenance. (Thaslima, J.S. et al, 2023).

   Data on the prevalence of root caries among Egyptian seniors are scarce and are mostly grey literature, which makes this data hard to find. The last published report for the prevalence of caries among Egyptian adults was carried out by the World Health Organisation (WHO) in collaboration with the Egyptian Ministry of Health in 2014. Therefore, the current study was carried out to investigate the prevalence of root caries among Egyptian seniors taking antihypertensive drugs in correlation with different risk factors. (Marwa M.S. Abbass et al,2019).
3. Rationale:

   Seniors age group are becoming the focus of attention in the dental community health approaches. They struggle with lower self-care ability and systemic health conditions such as hypertension. Hypertension and use of anti- hypertensive drugs has a definitive effect on pH levels of stimulated saliva which can be attributed to many oral detrimental changes such as xerostomia and dental caries. According to systematic reviews, around 50% of Egyptians over the age of 60 years old have hypertension. Also, among elderly, around 42% have a prevalence of dental caries and in 25 cross-sectional studies, 16 (64%) found positive correlation between age and root caries. (Hasan, M.D. et al,2014).

   Therefore, it is concluded that prevalence of root caries increases with age and it is greater in the elderly population than in younger adults. Therefore, old age can be a predictor of root caries since geriatrics usually have more gingival recession which leads to plaque accumulation and increase the risk of having root caries on exposed tooth root surfaces.

   Researchers believe that numerous hypertensive drugs have the capability to cause adverse effects in the oral cavity such as xerostomia and dental root caries but the association is still unclear. Also, it's not determined whether there are associated risk indicators or if they correlate with the pH levels of stimulated and unstimulated saliva.

   This study may help raise awareness among dentists and oral health care providers about dental health and its relation to antihypertensive drugs, also their possible side effects among seniors in Egypt. It aims to improve diagnosis and treatment plans, promote attention for seniors under a community health approach and educate different community members. The questionnaire will help evaluate the individual factors on patient's caries risk. Patients will be able to understand importance of regular dental examinations, the use of empirical therapy that can play a significant role in improving patient's quality of life and to consider oral health as a health issue to have a good perception of their oral health problem.
4. External Validity:

   1. This study could be generalised as the Faculty of Dentistry at Cairo University is considered a pivotal institution in Cairo governorates.
   2. The root (R) ICDAS assessment of caries lesions (Neeraj Gugnani et al., 2010) and the questionnaire (ICDAS root/coronal caries and individual factors in institutionalised elderly, Margarita Usuga-Vacca et al., 2021) are validated tools that have been used previously to assess the prevalence of carious lesions and associated risk indicators.
   3. Validation of the questionnaire:

      * The used questionnaire is validated because as it is designed similarly to the one used in a previously conducted cross-sectional study (Usuga-Vacca, M. et al., 2021).
5. Study design:

   1. Type of Study:

      * Analytical Cross- sectional study.
   2. Population:

      * Senior patients, age group of 50-70 years old attending Diagnostic Central Clinic at Cairo University Dental Educational Hospital.
   3. Exposure:

      * Anti- hypertension drugs.
   4. Setting:

      * This study will take place in postgraduate clinic Conservative Dentistry Department, Faculty of Dentistry, Cairo University.
6. Method of selection:

   * Seniors attending in the diagnosis clinic at Conservative Dentistry department, faculty of dentistry, Cairo University Egypt, will be examined for their chief complaint.
   * Patients will be enrolled in this study if they are compatible with eligibility criteria

ELIGIBILITY:
Inclusion Criteria:

* Senior patients, age group of 50-70 years old
* Positive subject acceptance for participation in the study
* Taking anti-hypertensive drugs
* Both gender
* Egyptian Nationals

Exclusion Criteria:

* Seniors with dental emergency 12
* Seniors with psychological problem
* Seniors with reported terminal illness or severe mental impairment in the medical records.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Senior patients, age group of 50-70 years old , attending in the diagnosis clinic at Conservative Dentistry department, faculty of dentistry, Cairo University Egypt, will be examined for their chief complaint.
  * Patients will be enrolled in this study if they are compatible with eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of root caries in patients taking anti- hypertensive drugs. | 3 months
  1. Prevalence of root caries measured by using the index of the root (R) 'ICDAS' assessment of caries lesions: Facial, mesial, distal, Lingual root surfaces of each tooth as one score/surface (decayed /filled) and its codes.
  2. Unit of measurement is:
     * Score E and 0 will be considered as root caries free and the rest of scores will be counted as root caries, Scores expressed as frequency and Percentages.
  3. The instrument used is: The root (R) ICDAS assessment of caries lesions using "Community Periodontal Index (CPI) probe", [WHO, 1997] with 0.5mm round tip.
  4. Participants included: All participants under inclusion criteria.

SECONDARY OUTCOMES:
Associated risk indicator | 4 months
  Associated risk indicators for all participants and Salivary assessment regarding pH level for each subgroup diagnosed with root caries lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumara-Raja B, Radha G. Prevalence of root caries among elders living in residential homes of Bengaluru city, India. J Clin Exp Dent. 2016 Jul 1;8(3):e260-7. doi: 10.4317/jced.52682. eCollection 2016 Jul. PMID 27398175
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] Langari SF, Hosseini SR, Bijani A, Jenabian N, Motalebnejad M, Mahmoodi E, Madani ZS, Sayadi F, Naghibi Sistani M, Ghadimi R, Baladi F, Hajimirzamohammad M, Mehryari M, Shirzad A. Association between antihypertensive drugs and the elderly's oral health- related quality of life: Results of Amirkola cohort study. Caspian J Intern Med. 2022 Summer;13(3):582-588. doi: 10.22088/cjim.13.3.582. PMID 35974945
- [Background] Valtellini R, Ouanounou A. Management of the Hypertensive Dental Patient. J Can Dent Assoc. 2023 Mar;89:n2. PMID 37098279
- See also: Biostatistics 102: quantitative data--parametric & non-parametric tests — https://pubmed.ncbi.nlm.nih.gov/14700417/
- See also: Streckfus CF, Strahl RC, Welsh S. Anti-hypertension medications: an epidemiological factor in the prevalence of root decay among geriatric patients suffering from hypertension. Clinical Preventive Dentistry. 1990 Aug-Sep;12(3):26-29. PMID: 2150630. — https://europepmc.org/article/med/2150630
- See also: Jingyang Zhang, Edward Chin Lo et al, (2020), Epidemiology of dental root caries: a review of risk factors, FOMM J. — https://fomm.amegroups.org/article/view/37409/html
- See also: Al-Harthy, N. , Qutiesha, A. et al, (2023) : A Preventive Strategy against Root Caries for the General Dentist: A Cross-sectional Clinical Study.Op Dent J, Volume 17. — https://opendentistryjournal.com/VOLUME/17/ELOCATOR/e187421062307310/FULLTEXT/